CLINICAL TRIAL: NCT03972683
Title: Novel Role of Acetylcholine in Regulating Vascular Tone: Effects of Age and Exercise Training
Brief Title: Role of Acetylcholine in Blood Flow Regulation in Healthy Adults: Effects of Age and Exercise Training
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Frank Dinenno, Professor, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACh sympatholysis
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Vasoconstriction; Vasodilation
Keywords: Exercise
MeSH Terms: conditions — Aneurysm; Motor Activity | interventions — Acetylcholine; Adenosine Triphosphate; Atropine; Phenylephrine; Nitroprusside

STUDY DESIGN:
Intervention Model Description: All participants will be studied before and after a handgrip exercise training intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Handgrip Exercise Training Intervention (Experimental): Participants will visit the lab for baseline measurements designed to evaluate signaling mechanisms that regulate blood flow. A physician will place a catheter in the brachial artery for pharmacological infusions. The following drugs will be administered to each participant: acetylcholine, adenosine triphosphate, atropine, phenylephrine, and sodium nitroprusside (see Interventions for further details regarding each drug). The order of infusions will be randomized and blood flow will be allowed to return to baseline between each infusion (~15 min) with the exception of atropine, which will be administered last owing to its longer half-life.
  Following baseline measurements, participants will complete a 7 week handgrip exercise training intervention, then they will return to the laboratory for post-training measurements. The post-training assessments will be performed in the same manner as the baseline visit; thus, the same drugs will be infused as described above.
  Interventions: Other: Handgrip Exercise Training; Drug: Acetylcholine; Drug: Adenosine Triphosphate; Drug: Atropine; Drug: Phenylephrine; Drug: Sodium Nitroprusside

INTERVENTIONS:
Other: Handgrip Exercise Training — Signaling mechanisms that regulate blood flow will be studied before and after 7 weeks of handgrip exercise training with the non-dominant forearm. Training sessions will consist of 30 min of rhythmic contractions using a handgrip exercise device, and participants will complete four training sessions per week.
Drug: Acetylcholine — Vasodilatory sensitivity to acetylcholine will be assessed in dose-response fashion as a standard test of vascular function. Doses of 0.5, 1.5, and 15 μg/dl forearm volume/min will be infused via a brachial artery catheter for 4 min per dose.
  Other Names: ACh
Drug: Adenosine Triphosphate — Vasodilatory sensitivity to adenosine triphosphate will be assessed during infusion of a dose of 10 μg/dl forearm volume/min administered via a brachial artery catheter over a total of 4 min.
  Other Names: ATP
Drug: Atropine — Atropine will be used to inhibit muscarinic acetylcholine receptors in order to determine the contribution of acetylcholine to vasodilation during exercise. An initial dose of 0.2 mg will be infused via a brachial artery catheter over 3 min, then a maintenance dose of 0.067 mg will be infused over 1 min prior to each of 5 subsequent experimental trials.
  Other Names: Atropine Sulfate
Drug: Phenylephrine — Vasoconstriction to phenylephrine will be used to assess sensitivity to alpha 1 adrenergic stimulation. Phenylephrine will be infused via a brachial artery catheter at 0.125 or 0.25 μg/dl forearm volume/min (18-35 and 60-85 age groups, respectively), adjusted according to forearm blood flow, for a total of 16 min.
  Other Names: Phenylephrine Hydrochloride
Drug: Sodium Nitroprusside — Sodium nitroprusside will be infused via a brachial artery catheter as a control vasodilator to elevate resting forearm blood flow to a level similar to that during exercise. The dose will be adjusted to match forearm blood flow to a similar level as during handgrip exercise, with an anticipated average dose of 1 μg/dl forearm volume/min. The dose will be infused for a total of 14 min.
  Other Names: SNP

SUMMARY:
The overall goal of this study is to address fundamental questions regarding how the molecule acetylcholine interacts with the sympathetic nervous system to regulate blood flow and oxygen delivery to working skeletal muscle in young and older adults. With advancing age, blood vessels supplying active muscle lose their ability to override sympathetic constriction, which limits delivery of oxygen and results in fatigue. Findings from these studies will serve as the foundation for new strategies to improve regional blood flow regulation in older adults and clinical populations, which will increase quality of life and help to preserve functional independence.

DETAILED DESCRIPTION:
The ability of blood vessels to dilate is essential to ensure adequate blood flow and oxygen delivery to active muscle during exercise. With advancing age, exercising muscle loses the ability to overcome vasoconstriction from the sympathetic nervous system, which impairs blood flow and limits exercise tolerance. Thus, understanding the signaling mechanisms that underlie the ability of active muscle to limit sympathetic vasoconstriction will advance our understanding of blood flow regulation in humans and lay the foundation for new strategies to improve blood flow and exercise tolerance in aging and clinical populations.

Therefore, the purpose of this research is to investigate endogenous acetylcholine as an important signaling molecule that regulates blood flow during exercise. The studies will also determine whether a reduced contribution of acetylcholine explains blood flow impairments in older adults. Since exercise training is known to improve acetylcholine signaling, this research will also address whether a handgrip exercise training intervention will improve blood flow regulation. The expected outcomes will provide new insight to the basic physiology underlying vascular control in humans. Furthermore, the findings will provide insight to the age-related decline in blood flow regulation during exercise and will assess the use of an exercise intervention to improve functional outcomes in older individuals.

Participants will be asked to complete several study visits over the course of 8 weeks. Once study eligibility has been determined, participants will report to the Human Performance Clinical Research Laboratory at Colorado State University for a 3 hour visit to assess forearm exercise capacity. In a separate 5 hour visit following an overnight fast, a physician will place a catheter in the brachial artery of the non-dominant arm to assess vascular function. Participants will then complete 7 weeks of handgrip exercise training (four sessions per week) and return to the laboratory for follow-up visits to assess forearm exercise capacity and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 OR 60-85

Exclusion Criteria:

* recent history of smoking
* body mass index greater than 30
* history of cardiovascular or metabolic disease, including hypertension or diabetes
* medications that may affect outcome measures, such as blood pressure medications or hormone replacement therapy
* high levels of exercise training, particularly with the forearm (such as weightlifting or rock-climbing)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional sympatholysis | Baseline (week 0) and post-intervention (week 8)
  Change in sensitivity to phenylephrine during handgrip exercise compared to rest

SECONDARY OUTCOMES:
Flow-mediated dilation | Baseline (week 0), mid-intervention (week 4), and post-intervention (week 8)
  Change in brachial artery diameter in response to increased shear rate

CONTACTS AND LOCATIONS:
Overall Officials: Frank Dinenno, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No